CLINICAL TRIAL: NCT04355169
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of Naldemedine in Patients Undergoing Surgeries That Include a Bowel Resection or Bowel Transection
Brief Title: A Study of Naldemedine in Participants Undergoing Surgeries That Include a Bowel Resection or Bowel Transection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated before the planned sample size was enrolled due to very slow enrollment.
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1902G1721
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Results first posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2021-12

CONDITIONS: Postoperative Gastrointestinal Dysfunction
Keywords: Bowel resection; Gastrointestinal recovery; peripherally acting mu-opioid receptor antagonist; Bowel transection
MeSH Terms: interventions — naldemedine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Naldemedine 1.25 mg (Experimental): Participants will receive 1.25 milligrams (mg) naldemedine twice daily (BID) beginning on the day of surgery (Day 1) and for up to a maximum of 10 days post-surgery.
  Interventions: Drug: Naldemedine
- Naldemedine 2.5 mg (Experimental): Participants will receive 2.5 mg naldemedine BID beginning on the day of surgery (Day 1) and for up to a maximum of 10 days post-surgery.
  Interventions: Drug: Naldemedine
- Naldemedine 5 mg (Experimental): Participants will receive 5 mg naldemedine BID beginning on the day of surgery (Day 1) and for up to a maximum of 10 days post-surgery.
  Interventions: Drug: Naldemedine
- Placebo (Placebo Comparator): Participants will receive matching placebo BID beginning on the day of surgery (Day 1) and for up to a maximum of 10 days post-surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naldemedine — Oral tablet
  Other Names: S-297995
  Arms: Naldemedine 1.25 mg; Naldemedine 2.5 mg; Naldemedine 5 mg
Drug: Placebo — Oral tablet
  Arms: Placebo

SUMMARY:
The objective of this study is to compare the efficacy of naldemedine versus placebo and to assess its effect on the time to gastrointestinal (GI) recovery following surgeries that include bowel resection and bowel transection.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo 1 of the following procedures via open (nonlaparoscopic) surgery under general anesthesia:

  * partial small or large bowel resection with primary anastomosis
  * radical cystectomy requiring bowel transection with primary anastomosis
* Planned to be managed postoperatively with an enhanced recovery protocol, which, at a minimum, includes all of the following elements:

  * early removal of the nasogastric tube, which is defined as removal of the nasogastric tube at the end of surgery
  * early ambulation, which is defined as ambulation on Day 1
  * early diet advancement on Day 1
* Planned to receive primary postoperative pain management with opioid analgesia administered by any route.
* American Society of Anesthesiologists (ASA) Physical Status Score of I, II, or III (a normal healthy participant, a participant with mild systemic disease, and a participant with systemic disease, respectively).

Exclusion Criteria:

* Scheduled to undergo a total colectomy or any procedure that results in a colostomy or ileostomy.
* Scheduled for endoscopic or laparoscopic surgery.
* Complete bowel obstruction.
* Complicated inflammatory bowel disease (such as ulcerative colitis or Crohn's disease).
* More than 2 major abdominal surgery (for example, gastrectomy, gastric bypass, gastric sleeve, lap banding, pancreatic resection, hepatectomy, intestinal transplant).
* More than 3 doses of an opioid (regardless of the route of administration) during the 7 days prior to surgery.
* Pregnancy or lactation.
* Presence of peritoneal catheter (for example, for dialysis or chemotherapy).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (8):
- United States (8):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Norton Hospital, Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - University of Louisville Division of Surgery, Louisville, Kentucky
  - Houston Methodist Hospital, Houston, Texas
  - CHRISTUS Mother Frances Hospital - Tyler, Tyler, Texas
  - CHRISTUS Trinity Clinic Research, Tyler, Texas
  - CHRISTUS Trinity Clinic Surgical Oncology, Tyler, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was terminated by the Sponsor. The Sponsor terminated the study based on the assessment that an adequate number of study sites were not able to reach the planned enrollment. Due to study termination and only 2 participants being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.
Groups:
- Naldemedine 1.25 mg: Participants received 1.25 milligrams (mg) naldemedine twice daily (BID) beginning on the day of surgery (Day 1) and for up to a maximum of 10 days post-surgery.
- Naldemedine 2.5 mg: Participants received 2.5 mg naldemedine BID beginning on the day of surgery (Day 1) and for up to a maximum of 10 days post-surgery.
- Naldemedine 5 mg: Participants received 5 mg naldemedine BID beginning on the day of surgery (Day 1) and for up to a maximum of 10 days post-surgery.
- Placebo: Participants received matching placebo BID beginning on the day of surgery (Day 1) and for up to a maximum of 10 days post-surgery.
Period: Overall Study
Arm/Group | Naldemedine 1.25 mg | Naldemedine 2.5 mg | Naldemedine 5 mg | Placebo
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study was terminated by the Sponsor. Due to study termination and only 2 participants being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.
Groups:
- Naldemedine 1.25 mg: Participants received 1.25 mg naldemedine BID beginning on the day of surgery and for up to a maximum of 10 days post-surgery.
- Naldemedine 2.5 mg: Participants received 2.5 mg naldemedine BID beginning on the day of surgery and for up to a maximum of 10 days post-surgery.
- Naldemedine 5 mg: Participants received 5 mg naldemedine BID beginning on the day of surgery and for up to a maximum of 10 days post-surgery.
- Placebo: Participants received matching placebo BID beginning on the day of surgery and for up to a maximum of 10 days post-surgery.
- Total: Total of all reporting groups
Arm/Group | Naldemedine 1.25 mg | Naldemedine 2.5 mg | Naldemedine 5 mg | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
Age, Continuous [unit: Years]
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Time From the End of Surgery to Time to First Toleration of Solid Food and First Bowel Movement (GI2)
Time Frame: Up to 10 days After Surgery
Population: as for baseline characteristics
Arm/Group | Naldemedine 1.25 mg | Naldemedine 2.5 mg | Naldemedine 5 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Time From the End of Surgery to Time When the Discharge Order is Written
Time Frame: Up to 10 days After Surgery
Population: as for baseline characteristics
Arm/Group | Naldemedine 1.25 mg | Naldemedine 2.5 mg | Naldemedine 5 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants Requiring Postoperative Reinsertion of the Nasogastric Tube
Time Frame: Up to 10 days After Surgery
Population: as for baseline characteristics
Arm/Group | Naldemedine 1.25 mg | Naldemedine 2.5 mg | Naldemedine 5 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants With Nausea on Days 1 Through 3
Time Frame: Days 1 to 3 After Surgery
Population: as for baseline characteristics
Arm/Group | Naldemedine 1.25 mg | Naldemedine 2.5 mg | Naldemedine 5 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants With Vomiting on Days 1 Through 3
Time Frame: Days 1 to 3 After Surgery
Population: as for baseline characteristics
Arm/Group | Naldemedine 1.25 mg | Naldemedine 2.5 mg | Naldemedine 5 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants Discharged by Day 10 Who Are Readmitted for Any Reason Within 30 Days After Discharge From the Hospital
Time Frame: From the Discharge Date (Days 1-10) up to 30 Days After Discharge
Population: as for baseline characteristics
Arm/Group | Naldemedine 1.25 mg | Naldemedine 2.5 mg | Naldemedine 5 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: This study was terminated by the Sponsor. Due to study termination and only 2 participants being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.
Description: This study was terminated by the Sponsor. Due to study termination and only 2 participants being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.
Arm/Group | Naldemedine 1.25 mg | Naldemedine 2.5 mg | Naldemedine 5 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study was terminated by the Sponsor. Due to study termination and only 2 participants being enrolled there are concerns regarding participant confidentiality, therefore no data are being reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PIs center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication.Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 45 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT04355169/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/69/NCT04355169/SAP_001.pdf